CLINICAL TRIAL: NCT05991375
Title: A Randomized Comparative Evaluation Of The Effects Of Dexmedetomidine As An Adjuvant With Bupivacaine In Supraclavicular Block In Chronic Renal Failure Patients Undergoing Basilic Vein Transposition Surgery
Brief Title: Comparison of Efficacy of Bupivacaine in Supraclavicular Block With or Without Dexmedetomidine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Syed Muhammad Abbas, Associate Professor, Department of Anaesthesia, Sindh Institute of Urology and Transplantation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIUT-ERC-2020/PA-257
Record Dates: First submitted 2023-07-29; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BUPIvacaine 0.25% (Active Comparator): (Injection bupivacaine (0.25%) 28 ml plus 2 ml. normal saline) making a total volume of local anaesthetic solution equal to 30 mL
  Interventions: Other: saline
- Bupivacaine0.25%+DEX (Experimental): Injection bupivacaine (0.25%) 28 mL plus dexmedetomidine I ug/kg diluted to 2 ml) making a total volume of local anaesthetic solution equal to 30 mL
  Interventions: Drug: DEXmedetomidine

INTERVENTIONS:
Drug: DEXmedetomidine — 28 mL of Bupivacain 0.25% was mixed with Dexmedetomidine 1 microgram/kg body weight mixed in 2 mL = total volume 30 mL
  Other Names: DEX
  Arms: Bupivacaine0.25%+DEX
Other: saline — 28 mL of Bupivacain 0.25% was mixed with 2 mL of Normal saline = total volume 30 mL
  Arms: BUPIvacaine 0.25%

SUMMARY:
End-stage renal disease (ESRD) patients are coming for Brachial vein transposition surgery. Patients were randomly allocated using sealed opaque envelope bearing A- (Injection bupivacaine (0.25%) 28 ml plus 2 ml. normal saline) and B-Injection bupivacaine (0.25%) 28 mL plus dexmedetomidine I ug/kg diluted to 2 ml).

Supraclavicular block under ultrasound and nerve stimulator guidance was performed.

DETAILED DESCRIPTION:
This study was conducted after approval of the institutional ethical review committee and then from College of Physicians and Surgeons Pakistan. Patients with end stage renal disease (ESRD) coming for Brachial vein transposition surgery, and fulfilling the inclusion criteria were enrolled in this study. All patients were instructed not to consume solid food after midnight prior to surgery. A brief history of demographic data was taken from each patient. Each participant's height in meters was measured using wall mounted scale, weight in kg using a weighing machine, and BMI kg/m² was noted prior to operation. The findings of quantitative variables (age, height, weight, sensory blockade, motor blockade and qualitative variables (gender, diabetes mellitus type II, hypertension, and dyslipidemia) were entered in the proforma attached as an annexure. Patients were randomly allocated using sealed opaque envelope bearing A- (Injection bupivacaine (0.25%) 28 ml plus 2 ml. normal saline) and B-Injection bupivacaine (0.25%) 28 mL plus dexmedetomidine I ug/kg diluted to 2 ml). Only the anaesthesiologists for the specific case were aware of the treatment allocation until the end of the surgical procedure. The investigator for assessing the block and the other outcome variables, remained blinded to the patient's group allocation.

Routine monitoring of heart rate & rhythm by ECG, and arterial blood pressure using non-invasive blood pressure (NIBP) including systolic, diastolic & mean arterial blood pressure, and peripheral oxygen saturation (SPO2) using a pulse oximeter was performed on each patient. The supraclavicular brachial plexus block was performed under the supervision of a consultant anaesthesiologist in a supine position with a head up to 45 degrees. An Intravenous (IV) line was established and the skin was disinfected and a linear probe, high frequency 12 MHz was placed firmly over the supraclavicular fossa, the probe was positioned in the transverse plane immediately superior to the clavicle at approximately its midpoint. The probe was tilted caudally to obtain a cross sectional view of the subclavian artery. The brachial plexus was seen as a collection of hypo-echoic oval structures lateral and superficial to the artery. Using a 25 gauge needle 1 to 2 ml of 2% lidocaine was locally infiltrated into the skin 1 cm lateral to the probe to decrease the discomfort during needle insertion. A 50 mm or 80 mm length, short bevel, insulated nerve stimulator needle was used. Peripheral nerve stimulation (PNS) is an additional way of confirming nerve location. Initial settings was set at 0.5 mA current, 2 Hz frequency, and pulse width of 0.1 milliseconds. Close approximation to the divisions of brachial plexus was confirmed by getting nerve stimulation on 0.3 mA current. The needle was advanced along the long axis in the same plane as the ultrasound beam. The shaft and tip was visualized in real time as the needle was advanced towards the target nerves. The drug in either group was injected under direct vision of ultrasound beams and by confirming with nerve stimulation. Sensory blockade and motor blockade was assessed every 3 minutes. Time of onset of sensory and motor blockade and duration of sensory and motor blockade were noted as per operational definition. Postoperative pain was assessed with visual analogue scale (VAS). Patients were asked to mark a point on the line that matches the intensity of pain on the Visual Analogue Score hourly for 4 hours post operatively. Those patients having arm pain equal to or greater than 4 on VAS, were given rescue analgesic (inj. Paracetamol (15mg/kg 1/V) and duration of analgesia were noted as per operational definition.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure patients who will undergo elective basilic vein transposition surgery
* Either gender
* ASA III
* Age 18-65 years.

Exclusion Criteria:

* Mentally challenged
* Pregnancy.
* Hypersensitivity to bupivacaine or dexmedetomidine
* Seizures
* Neck swelling (hematoma, lipoma, tumor, thyroid)
* Neuromuscular dystrophy
* Bleeding disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Pain score | 0-4 hours
  Visual Analogue Scale for pain
  0-1-2-3-4-5-6-7-8-9-10
  Pain score 0 means no pain, Pain score 1 to 3 means mild pain, Pain score 4-6 means moderate pain, Pain score 7-9 means severe pain, Pain score 10 means most excruciating pain one can have,
Heart rate | 0-4 hours
  Heart rate as per vitals monitoring device
Mean blood pressure | 0-4 hours
  as measured by non-invasive blood pressure monitoring device

CONTACTS AND LOCATIONS:
Overall Officials: Fauzia Ali, FCPS, Study Chair — Professor Dept of Anaesthesiology
Locations (1):
- Syed Muhammad Abbas, Karachi, Sindh, Pakistan